CLINICAL TRIAL: NCT03084029
Title: The Neural Basis of Oxytocin's Effects on Empathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, PhD, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-03
Record Dates: First submitted 2016-04-15; First posted 2017-03-20 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: oxytocin; fMRI; empathy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- male participants - oxytocin nasal spray (Experimental): male participants - receiving a single dose of 40 IU intranasal oxytocin
  Interventions: Drug: Oxytocin
- female participants - oxytocin nasal spray (Experimental): female participants - receiving a single dose of 40 IU intranasal oxytocin
  Interventions: Drug: Oxytocin
- male participants - placebo nasal spray (Placebo Comparator): male participants - receiving a single dose of 40 IU intranasal placebo
  Interventions: Drug: Placebo
- female participants - placebo nasal spray (Placebo Comparator): female participants - receiving a single dose of 40 IU intranasal placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 international units
  Other Names: Oxytocin Treatment
  Arms: female participants - oxytocin nasal spray; male participants - oxytocin nasal spray
Drug: Placebo — 40 international units
  Other Names: Placebo treatment
  Arms: female participants - placebo nasal spray; male participants - placebo nasal spray

SUMMARY:
The main focus of this study is to examine oxytocin effects on behavioral and neural indices of empathy processing.

DETAILED DESCRIPTION:
The neuropeptide oxytocin (OXT) has been demonstrated to modulate empathy in previous behavioural studies. The present study aims at replicating previous findings on OXT on empathy as well as to determine the neural basis of these effects.

In a between-subject, randomized double-blind design, subjects will be either administered intranasal OXT or placebo nasal spray (40 IU). 45 minutes after administration subjects will undergo (fMRI) tasks of empathic processing.

During the tasks subjects will be shown empathy inducing stimuli, and the behavioral and neural response in terms of cognitive, emotional and indirect emotional empathy will be assessed.

Before the administration of treatment, validated questionnaires assessing potential confounding variables, such as depression (Becks Depression Inventory (BDI)) or mood (Positive And Negative Affect Scale (PANAS)) will be administered to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* no smoking at least 12 hours before experiment
* no alcohol, coffee or other stimulant drinking at least 12 hours before experiment

Exclusion Criteria:

* mental implants
* pregnancy
* uterine cavity operations
* use of medication
* acute physical disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Neural processing of empathy as assessed using fMRI | 45-115 minutes after single dose administration
  Main effects of treatment and interaction between treatment effects and sex will be assessed on brain activity and connectivity in core regions of the empathy networks during processing of empathy inducing pictures

SECONDARY OUTCOMES:
Behavioral ratings of subjective experienced empathy processing | 45-115 minutes after single dose administration
  Main effects of treatment and interaction between treatment effects and sex will be assessed on subjective feelings of empathy (ratings on a Likert scale in response to empathy inducing pictures).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — China,Sichuan, School of Life Science and Technology,University of Electronic Science and Technology
Locations (1):
- School of Life Science and Technology,University of Electronic Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No